CLINICAL TRIAL: NCT03357185
Title: Prospective Evaluation of Femoral Tripod Eversion Technique
Acronym: Eversion
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD0515
Record Dates: First submitted 2017-11-24; First posted 2017-11-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Atheromatous
Keywords: Femoral bifurcation; Peripheral arterial disease; Vascular surgery; Eversion; Open surgery
MeSH Terms: conditions — Plaque, Atherosclerotic; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Femoral eversion — The purpose of this database is to compile the data of patients followed at the René Dubos Hospital Center with symptomatic lower extremity arterial disease (AOMI) (Rutherford 2 to 5) who were operated on by the femoral tripod eversion technique.
  The database will include data on the operation, possible complications, clinical course of patients and medical and surgical follow-up.

SUMMARY:
Endarteriectomy is considered as the first line treatment of femoral bifurcation atheromatous lesions. Eversion technique, similar to that used for carotid bifurcation, is safe and possible for the majority of the femoral tripod lesions. The major advantage of the eversion technique is the absence of prosthetic material to be performed. However, its use has been scarcely evaluated in the literature to date. This work aims at evaluating the long term safety and the efficacy of eversion femoral technique. Surgical technique was thoroughly described and participants were followed up for two years by serial clinical and doppler US examination.

DETAILED DESCRIPTION:
Femoral bifurcation lesions is one of the most frequent lesion encountered in lower limb atheromatous occlusive disease. Current treatment options consists in femoral endarteriectomy or bypass. More recently, endovascular treatment of femoral tripod lesions has been reported. Inguinal area is prone to postoperative infection in up to 20% of the cases. Hence, the use of synthetic graft puts the participants at risk of dramatic consequences in case of postoperative infection. Besides, long term data are still required to validate the use of endovascular device in this very "surgical" area. The use of the eversion technique is possible in the majority of the lesions and offer the major advantage of open surgery in terms of durability, without the use of synthetic material in case of postoperative infection.

The investigators herein report the detailed technique, tips and variations of the eversion technique as well as the clinical follow up in terms of clinical benefit according to Rutherford classification and restenosis evaluated by serial doppler US.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Lower limb atheromatous occlusive disease.
* Stage 2 to 4 according to Rutherford's classification

Exclusion Criteria:

* Age< 18
* Previous surgery or endovascular treatment of the ipsilateral limb
* Non atheromatous disease
* Pregnancy
* Life-expectancy estimated to be less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Register including all patients who have been treated with the femoral eversion technique.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Clinical follow-up | One year.
  Observation of the clinical and life-threatening status of the participants twelve months after the operation. From a general point of view observation of clinical improvement according to Rutherford classification.

SECONDARY OUTCOMES:
Clinical complications | At one month, six months and twelve months.
  Clinical follow-up and echo-Doppler was obtained at one month, six months and twelve months.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel DAVAINE, Principal Investigator — Hôpital NOVO

IPD SHARING:
Plan to Share IPD: No